CLINICAL TRIAL: NCT02100800
Title: Assessment of Emphysema in COPD Patients Using 1.5T MR Imaging With Ultrashort Echo Time (UTE) Pulse Sequences
Brief Title: Assessment of Emphysema Using 1.5T MRI With UTE Pulse Sequences
Acronym: EMPHYREM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHUBX 2012/09; 2013-A00353-42 (Other: ANSM)
Record Dates: First submitted 2014-03-18; First posted 2014-04-01 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Emphysema
Keywords: COPD; Emphysema; MRI; UTE; Quantification; CT
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- COPD Group (Experimental): 30 patients with diagnosis of COPD
  Interventions: Other: MR and CT measurements of emphysema quantification
- Control Group (Sham Comparator): 10 volunteers with extrapulmonary neoplasia
  Interventions: Other: MR and CT measurements of emphysema quantification

INTERVENTIONS:
Other: MR and CT measurements of emphysema quantification

SUMMARY:
Emphysema is a major pathological feature of Chronic Obstructive Pulmonary Disease (COPD). Non-invasive assessment of emphysema is a crucial issue for the phenotype and follow-up of COPD patients. Currently, CT is the method of reference to evaluate and quantify emphysema but it remains a radiation-based technique. Magnetic Resonance Imagery (MRI) with ultrashort echo time (UTE) pulse sequences is a promising non-ionizing alternative for lung imaging. Our objective is to evaluate emphysema in COPD patients using CT and MR-UTE, and to test the agreement between both techniques.

DETAILED DESCRIPTION:
COPD is a major public health problem and is pathologically characterized by lung emphysema and bronchial remodeling. Emphysema is defined as an irreversible destruction of alveolar walls and subsequent enlargement of air spaces. New targeted therapies against emphysema are currently developed, thereby stressing the need for non-invasive tools aimed at quantifying emphysema. Multi-slice computed tomography (CT) is the method of reference to quantify emphysema but involves ionizing radiation, thus limiting the possibility of long-term follow-up. MRI is a non-ionizing 3D imaging technique; however, lung MRI is technically challenging with the result that it is currently not used in routine practice. Indeed, both low proton density and susceptibility effects lead to a very low signal intensity derived from lung parenchyma. Recently, pulse sequences with ultrashort echo time (UTE) have been implemented by the use of half radio-frequency excitations and radial projection reconstruction. These UTE sequences make it theoretically possible to retrieve more signal from the lung parenchyma. We aim at using 3D T1-weighted UTE pulse sequences on a 1.5T magnet (Avanto dot, Siemens) in COPD patients in order to distinguish normal lung from emphysematous areas. Thirty COPD patients and 10 volunteers are expected to take part in the study. All will benefit from Pulmonary Functional Testing (PFT), CT and MRI. Our strategy will consist in quantifying pulmonary emphysema using MRI and CT in those subjects, testing for correlations between MR and CT measurements and assessing the reproducibility of emphysema quantification using MRI. Our objective is to demonstrate that MR-UTE pulse sequence at 1.5T is accurate and reproducible in evaluating and quantifying pulmonary emphysema.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged more than 40 years.
* COPD group: patients with diagnosis of COPD at distance (minimum 4 weeks) from any acute exacerbation; staging 1-4 according to 2010 GOLD guidelines. PFTs and chest CT-scan should be available within a maximum of 30 days before inclusion.
* Control group: subjects without any chronic symptoms such as cough or expectoration (St-Georges symptoms scoring < 5%), with normal chest CT-scans performed in the pretherapeutic work-up of extrapulmonary cancers within a maximum of 30 days before inclusion. These subjects will be age- and sex-matched with COPD patients.
* With a written informed consent and health insurance.

Exclusion Criteria:

* Subjects without any social security or health insurance.
* History of asthma, lung fibrosis, pulmonary hypertension or cystic fibrosis.
* Pregnancy.
* Any respiratory treatment for control subjects.
* MRI contraindications: Magnetically activated implanted devices (cardiac pacemakers, insulin pumps, neurostimulators, cochlear implants), metal inside the eye or the brain (aneurysm clip, ocular foreign body), cardiac valvular prosthesis (Starr-Edwards pre-6000), subject with claustrophobia.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2016-07-13 (Actual); Study Completion 2016-07-13 (Actual)

PRIMARY OUTCOMES:
Agreement between MRI and CT for evaluating the regional distribution of emphysema | During MRI and CT, Day one
  MRI and CT evaluation of regional distribution of emphysema will be assessed by 2 blind radiologists. Agreement between both evaluation will be assessed during statistical analyses after study completion

SECONDARY OUTCOMES:
Agreement between MRI and CT for evaluating the presence of emphysema | During MRI and CT, Day one
  MRI and CT evaluation of presence of emphysema will be assessed by 2 blind radiologists. Agreement between both evaluations will be assessed during statistical analyses after study completion
Correlation between emphysema scoring extracted from CT and MR images | During MRI and CT, Day one
  Emphysema scoring will be assessed by 2 blind radiologists. Correlation between both evaluations will be assessed during statistical analyses after study completion
MR emphysema reproductibility scoring over the time | During MRI, Day one
  During MRI emphysema scoring will be assessed a second time after 10 minutes wait
Comparison of MR emphysema scoring and lung signal values between COPD and controls | During MRI, Day one
  MR emphysema scoring and lung signal values collected during MRI will be assessed during statistical analyses after study completion and compared between COPD and controls
Comparison of MR emphysema scoring between different GOLD stages | During MRI, Day one
  MR emphysema scoring collected during MRI will be assessed during statistical analyses after study completion and compared between different GOLD stages
Correlation between MR emphysema scoring and PFT obstructive indexes (FEV1, FEV1/FVC, DEMM25-75) | During MRI, Day one
  MR emphysema scoring and PFT obstructive indexes collected during MRI will be assessed during statistical analyses after study completion.
Comparison of signal-to-noise and contrast-to-noise ratios of lung parenchyma measured using UTE MRI and classical pulse sequences, as well as image quality assessed using a 4-point scale. | During MRI, Day one
  Signal-to-noise and contrast-to-noise ratios of lung parenchyma collected during MRI will be assessed during statistical analyses after study completion and compared between measures using UTE MRI and classical pulse sequences.

CONTACTS AND LOCATIONS:
Overall Officials: Gaël DOURNES, MD, Principal Investigator — University Hospital Bordeaux (France)
Locations (1):
- University Hospital Bordeaux, Pessac, France

REFERENCES:
- [Derived] Benlala I, Berger P, Girodet PO, Dromer C, Macey J, Laurent F, Dournes G. Automated Volumetric Quantification of Emphysema Severity by Using Ultrashort Echo Time MRI: Validation in Participants with Chronic Obstructive Pulmonary Disease. Radiology. 2019 Jul;292(1):216-225. doi: 10.1148/radiol.2019190052. Epub 2019 Jun 4. PMID 31161972